CLINICAL TRIAL: NCT01828359
Title: An Eight-week, Randomized, Double-blind Multicenter Study to Compare the Efficacy and Safety of Amosartan® Tab 5/100mg Versus Cozaar® Plus Pro Tab in Patients With Essential Hypertension Uncontrolled With Losartan 100mg Monotherapy
Brief Title: The Efficacy and Safety Study of Anti-hypertension Combination Drug in Patients Uncontrolled With Monotherapy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-ALOS-401
Record Dates: First submitted 2013-04-07; First posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan; Proline; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amosartan® tab (Experimental): Amlodipine 5mg /Losartan 100mg
  Interventions: Drug: Amosartan® tab
- Cozaar® plus pro tab (Active Comparator): Losartan 100mg/ HCTZ 12.5mg
  Interventions: Drug: Cozaar® plus pro tab

INTERVENTIONS:
Drug: Amosartan® tab — comparison of different combination of anti-hypertension drug
  Other Names: Amlodipine 5mg /Losartan 100mg
  Arms: Amosartan® tab
Drug: Cozaar® plus pro tab — comparison of different combination of anti-hypertension drug
  Other Names: Losartan 100mg/ HCTZ 12.5mg
  Arms: Cozaar® plus pro tab

SUMMARY:
The purpose of this study is to evaluate the blood pressure lowering effects of an amlodipine/losartan combination treatment and losartan/Hydrochlorothiazide combination treatment in patients with essential hypertension uncontrolled with losartan 100mg monotherapy.

DETAILED DESCRIPTION:
* Quality assurance plan was implemented by site monitoring, including data validation and registry procedures and Source data verification to assess the accuracy, completeness by comparing the data to external data sources (medical records and paper case report forms).
* Data dictionary contains the registry, including the source of the variable, coding information (MedDRA ver12.0), and normal ranges.
* Statistical analysis were performed using SAS® Version 9.2, SAS institute, Cary, NC, USA

ELIGIBILITY:
Inclusion Criteria:

* 20 aged or over
* Patients with blood pressure measured at Visit 1; 90mmHg≤MSDBP mmHg if on anti-hypertensive drugs, 95mmHg≤MSDBP mmHg if not on anti-hypertensive drugs
* Patients with blood pressure measured at Visit 2 were 90mmHg≤MSDBP mmHg (non-responder to Losartan 100mg for 4-week treatment)

Exclusion Criteria:

* Patients with too high Blood pressure

  •≥ sitSBP 20mmHg or ≥ sitDBP 10mmHg of variation in three measurements from the reference arm selected at Screening
* History of hypersensitivity to CCB ,Angiotensin II receptor blockers or Sulfonamide.
* Secondary hypertension or suspected to be

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Mean Sitting Diastolic Blood Pressure (MSDBP) | Baseline, Week 8

SECONDARY OUTCOMES:
Change from baseline in MSDBP | Baseline, week 4
Change from baseline Mean Seated Systolic Blood Pressure (MSSBP) | Baseline, Week 4 and 8
Blood pressure responder rate | Baseline, Week 4 and 8
  Rate of patients who achieved target blood pressure (MSSBP < 140 mmHg and MSDBP < 90 mmHg), or MSSBP decrease > 20 mmHg from baseline or MSDBP decrease > 10 mmHg from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Taehoon Ahn, Ph.D., Principal Investigator — Gachon University Gil Medical Center